CLINICAL TRIAL: NCT01961128
Title: Pilot Feasibility Study of the Use of Random Periareolar Fine Needle Aspiration Exercise Induced Changes in Breast Tissue
Brief Title: RPFNA Assessment of Exercise Effect in Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer A. Ligibel, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 11-291
Record Dates: First submitted 2013-01-04; First posted 2013-10-11 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Breast Cancer
Keywords: High risk
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Intervention (Experimental): 220 minutes of exercise per week, including 2-3 supervised sessions for 6 weeks
  Interventions: Behavioral: Exercise Intervention

INTERVENTIONS:
Behavioral: Exercise Intervention

SUMMARY:
This study is being done to see if the investigators can measure changes that occur in breast tissue when women at risk of developing breast cancer start an exercise program. The investigators are interested in studying this because research shows that women who exercise regularly are less likely to develop breast cancer, but there is not very much information explaining how exercise could affect breast cells in a way to prevent cancer from occurring. In this research study the investigators will use a research technique called breast random fine needle aspiration (RPFNA) to test breast cells for their shape and how they look. The investigators will look at breast cells before and after a participant takes part in an exercise program to see if the investigators are able to see any changes in breast cells that could have happened due to the exercise program. This research will help us to develop larger projects to see if exercise programs could be helpful in preventing breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* History of lobular carcinoma in situ, atypical ductal/lobular hyperplasia on prior breast biopsy or lifetime risk of breast cancer of at least 20% based on any risk model, or personal history of BRCA1 or 2 mutation
* Physically able to exercise and physician consent to start an exercise program
* Sedentary activity pattern
* Premenopausal
* English speaking and able to read English

Exclusion Criteria:

* History of invasive breast cancer or ductal carcinoma in situ
* Absolute contraindications to maximal exercise testing as recommended by the American Thoracic Society
* Any condition which in the investigator's opinion makes the subject unsuitable for study participation
* Participating in another clinical study with competing study outcomes
* Pregnant or breastfeeding
* Unable to comply with protocol and/or not available for follow-ups
* Type II Diabetes
* Allergic to local anesthetics
* History of bilateral or unilateral mastectomy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of enrolling patients in a study looking at the impact of exercise upon breast tissue markers | 2 years
  This is a small pilot feasability study designed to see if we can recruit patients into this kind of trial and if we can measure biomarker expression in breast tissue collected through RPFNA.
  Data analyses will be primarily descriptive in this pilot study. The primary feasibility endpoint will be assessed by the number of women with pre- and post-exercise RPFNA samples with sufficient cells (> 500) for analysis. We require evidence that at least 60% of participants could provide adequate samples order to declare success in this pilot study. Therefore, if 10 of 12 enrolled women have RPFNA samples at both times with sufficient cells, the lower bound of the one-sided, 90% exact confidence interval will exceed 60% and the study will be considered feasible.

SECONDARY OUTCOMES:
Secondary objectives will explore changes in proliferative and morphologic indices of the breast as expressed by changes in Ki-67 and the Masood index. | 2 years
  Baseline values of percent Ki-67 and Masood index will be summarized using descriptive statistics. The proportions of women with 6-week changes in Masood index of 0 points, 1-2 points, and 3 or more points will be summarized, as will changes in Ki-67 percent. Comparable analyses will be conducted to estimate the changes in concentrations of serum metabolic and inflammatory biomarkers: insulin, glucose, IGF-1, IGFBPs, IL-2, IL-6, CRP, and TNFα. We will also summarize changes in expression of metabolic, sex steroid and related receptors in epithelial breast tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ligibel, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States